CLINICAL TRIAL: NCT04229472
Title: Characterising the Stable and Dynamic Left Atrial Substrate in Atrial Fibrillation Using High Density Contact and Non-contact Mapping
Brief Title: Characterising the Stable and Dynamic Left Atrial Substrate in Atrial Fibrillation
Acronym: CASDAF-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Tim Betts MD MBChB FRCP, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14295
Record Dates: First submitted 2020-01-07; First posted 2020-01-18 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Normal subject control group (Experimental): High density mapping of left atrial voltages in patients with supraventricular tachycardia
  Interventions: Diagnostic Test: High density electrophysiological mapping
- Atrial fibrillation group (Experimental): High density mapping of left atrial voltages
  Interventions: Diagnostic Test: High density electrophysiological mapping
- AcQMap atrial fibrillation group (Experimental): High density mapping of left atrial voltages and AcQMap propagation patterns alongside cardiac MRI
  Interventions: Diagnostic Test: High density electrophysiological mapping; Diagnostic Test: Cardiac Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: High density electrophysiological mapping — Recording of electrophysiological data using a high density contact catheter during pacing at the time of catheter ablation for atrial fibrillation.
Diagnostic Test: Cardiac Magnetic Resonance Imaging — Late gadolinium enhance cardiac magnetic resonance imaging (in AcQMap group only)
  Arms: AcQMap atrial fibrillation group

SUMMARY:
Atrial fibrillation (AF) is the most common sustained arrhythmia, with increasing prevalence associated with an ageing population. Management is challenging, and invasive catheter ablation procedures are increasingly used in those with symptoms refractory to drug therapy. Unfortunately, success rates from this procedure can be limited. This is partly due to limitations in understanding of the mechanisms involved in arrhythmia propagation. There is much interest in the role of structural changes within the muscle of the left atrium resulting in scaring (known as fibrosis). This has been identified on MRI studies and invasive electroanatomical mapping using voltage amplitude of recorded signals as a surrogate measure of tissue properties. This however is affected by the technology used, as it does not routinely incorporate the effect of heart rate on conduction properties. Furthermore, although this aims to identify regions of structural changes, it does not identify more dynamic patterns of conduction seen during AF.

This study aims to use a high density mapping catheter (Abbott Advisa HD grid (SE)), which employs a novel algorithm to minimise the effect of wavefront direction on the size of electrical signals. Electroanatomical mapping of the left atrium in patients with atrial fibrillation will be conducted whilst pacing at long and short cycle lengths to assess the effect of pacing rate on conduction properties, assessed using signal morphology and conduction velocity. The same procedure will also be carried out in 5 control patients to allow comparison with normal atria. Two subgroups will also analysed. In the first the aim is to compare the use of the HD grid catheter to a bipolar ablation catheter in carrying out electroanatomical mapping. In the second, to correlate electrical signals obtained with propagation patterns identified using the AcQMap non-contact mapping system and atrial properties identified on cardiac MRI.

DETAILED DESCRIPTION:
This is a prospective, non-randomised mechanistic study of 35 patients, including 5 control patients with normal atria and 30 patients with atrial fibrillation.

The 5 control patients will be undergoing an elective catheter ablation for another arrhythmia (likely supraventricular tachycardia (SVT)) involving a trans-septal puncture for left atrial access.

The 30 main study participants will only be patients who are already planning to undergo a catheter ablation procedure for atrial fibrillation. This will include 10 patients who are undergoing elective AcQMap guided procedures, in order to correlate non-contact propagation patterns with contact substrate mapping. These 10 patients will also undergo cardiac MRI imaging.

Study participants will be identified by medical staff in the outpatient clinic at the time of listing for catheter ablation, or by review of patients electronically listed for this procedure. If patients are in the clinic and give consent then a member of the research team may approach them at this stage. If identified by medical staff through listing for the procedure, they will be approached by telephone. An information leaflet will then be provided by post or email (if this has not been provided in clinic) with contact details for the research team. If willing to participate then formal screening and recruitment will take place at the time of attendance for standard pre-procedure assessment appointments or when attending for the elective procedure. Information must have been provided with sufficient time for the potential participant to fully consider involvement prior to formal recruitment and consent (generally expected to be at least 24 hours). It will be clear that participation or choosing not to participate has no impact on proceeding with their planned procedure. As the baseline assessments required involve purely a review of a participants medical history and measurement of height and weight, this will be combined with the screening/recruitment visit, and providing information has been provided sufficiently in advance then may be undertaken at the time of attending for the study procedure.

Study procedure:

In line with standard practice in this institution, all AF ablation procedures will be undertaken under general anaesthesia. SVT ablation will be conducted under sedation. Venous access, trans-septal puncture and placement of standard electrophysiology catheters will be undertaken in accordance with standard clinical care. Anticoagulation will be administered following trans-septal puncture in line with standard protocols.

All participants:

All study participants will undergo electroanatomical voltage mapping (EAVM) using the Abbott Advisa HD Grid (SE) mapping catheter using the orthogonal wave setting (HD wave solution). If in AF at the start of the procedure then direct current cardioversion (DCCV) will be used to restore sinus rhythm. This can be repeated at the discretion of the operator if initially unsuccessful (including internal cardioversion if necessary). If unsuccessful then the patient will no longer be included in the study. Mapping will then be undertaken during bipolar pacing from the mid point of the coronary sinus catheter whilst pacing at 800ms for 4 beats followed by a single beat at 300ms (or the shortest captured if longer). Ablation and the rest of the procedure can then be performed according to standard clinical practice.

For the 30 patients undergoing AF ablation, once the initial study procedures above are complete, further mapping will be conducted using either an ablation catheter (20 patients) or the AcQMap system (10 patients).

Ablation catheter mapping:

This involves using a contact force guided bipolar irrigated ablation catheter (Abbott Tacticath) during the same pacing protocol. For patients presenting in sinus rhythm or AF, all required mapping should be completed in the presenting rhythm followed by either AF induction (using incremental burst atrial pacing) or DCCV respectively before completion of mapping procedures. Ablation in line with standard clinical care will be undertaken following completion of all mapping procedures.

AcQMap guided mapping and ablation:

10 patients with persistent AF who are undergoing AcQMap guided elective catheter ablation procedures will be included. All patients will undergo the same main study mapping procedure outlined above. In addition, AcQMap recordings will also be obtained. Recordings will be made during pacing with the same main study protocol and two 30second recordings will be undertaken during AF. HD grid contact recordings will then also be obtained in regions of prominent rotational and irregular conduction identified by AcQMap and ablation performed at the operator's discretion.

Post procedure care including subsequent discharge will continue in line with standard clinical practice and no study follow up is required (excluding the repeat MRI referred to below).

Cardiac MRI:

The 10 participants undergoing elective AcQMap guided procedures will also undergo a cardiac MRI both prior to and after the procedure. The initial scan will be within the 6 weeks prior to the ablation procedure and the follow up scan will be within 3-6 months after the procedure. These will be planned whenever possible to take place alongside routine hospital visits.

Patients will complete an MRI safety questionnaire (5 minutes) prior to the scan. An intravenous cannula will be inserted. Cardiac MRI will evaluate cardiac structure and function, with particular focus on the left atrium. For late gadolinium enhancement imaging, the total dose of gadolinium-based contrast will not exceed 0.2mmol/kg.

The total duration of the MR protocol will be approximately 60 minutes, considering approximately 50 minutes of scanning time, plus approximately 10 minutes for pre/post-scan preparation.

It is planned that a total of 35 patients will be recruited to this study. As this study is not evaluating clinical outcomes of a procedure, greater numbers are not needed. This number is thought to be enough to reveal any patterns in electrophysiological properties. Data analysis will occur offline using anonymised datasets. Results will be collated and a report compiled at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with paroxysmal or persistent atrial fibrillation and planned for a catheter ablation procedure (AF ablation group only).
* Undergoing elective left sided catheter ablation procedure involving a trans-septal approach (Control group only).
* In the Investigator's opinion the participant is able and willing to comply with all trial requirements.

Exclusion Criteria:

* Previous cardiac surgery.
* Previous left atrial ablation (catheter or surgical).
* Medical history including any of: atrial fibrillation, atrial flutter, hypertension, diabetes mellitus, chronic obstructive pulmonary disease, significant mitral valve disease (stenosis or regurgitation), pulmonary hypertension, obstructive sleep apnoea, ischaemic heart disease, cerebrovascular disease, peripheral vascular disease, structural heart disease (excluding known accessory pathway), congenital cardiac anomaly (excluding accessory pathway), previous left atrial ablation (catheter or surgical), cardiac surgery (control group only).
* Contraindications to MR scanning (such as metallic or electronic objects implanted in your body or history of severe claustrophobia) (AcQMap guided ablation group).
* Significantly impaired renal function (eGFR<30ml/min).
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational medicinal product in the past 12 weeks. (Involvement in any other research trial is not a contraindication per se).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Betts, MD MBChB FRCP, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Subject Control Group | Atrial Fibrillation Group | AcQMap Atrial Fibrillation Group
Started | 0 | 20 | 11
Completed | 0 | 19 | 10
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Due to recruitment challenges during the COVID-19 pandemic, we were unable to enroll normal subjects as initially planned.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Subject Control Group | Atrial Fibrillation Group | AcQMap Atrial Fibrillation Group | Total
Number analyzed (Participants) | 0 | 19 | 10 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 5 | 4 | 9
  Male |  | 14 | 6 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Ablation Type [Count of Participants; unit: Participants]
  De novo |  | 19 | 6 | 25
  Redo |  | 0 | 4 | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] |  | 65 (10) | 64 (9) | 64 (10)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] |  | 30 (5) | 31 (5) | 30 (5)

OUTCOME MEASURES:

1. Primary Outcome: To Define the Normal Range of Voltage Amplitude
Description: Mean and distribution of left atrial voltage amplitude across the whole chamber and by segments with lower limit of normal defined as the upper 95% value within the segment with the lowest mean amplitude at long pacing cycle length.
Time Frame: During ablation procedure
Population: It was not possible to maintain sinus rhythm during recordings at long pacing cycle lengths in all patients.
Measure: Mean (Standard Deviation); unit: mV
Groups:
- AcQMap Atrial Fibrillation Group: High density mapping of left atrial voltages
Arm/Group | Atrial Fibrillation Group | AcQMap Atrial Fibrillation Group
Number analyzed (Participants) | 9 | 8
mV | 2.00 (2.39) | 1.92 (2.37)

2. Other Pre Specified Outcome: Evaluate the Effect of Cycle Length on Electrogram Morphology in Normal Subjects
Description: A change in electrogram morphology from normal to abnormal (defined as ≥3 deflections lasting ≥50ms), between long and short pacing cycle length.
Time Frame: During ablation procedure
Population: as for baseline characteristics
Arm/Group | Normal Subject Control Group | Atrial Fibrillation Group | AcQMap Atrial Fibrillation Group
Number analyzed (Participants) | 0 | 0 | 0

3. Other Pre Specified Outcome: Evaluate the Effect of Cycle Length on Electrogram Amplitude in Normal Subjects
Description: A change in electrogram voltage amplitude between long and short pacing cycle length.
Time Frame: During ablation procedure
Population: as for baseline characteristics
Arm/Group | Normal Subject Control Group | Atrial Fibrillation Group | AcQMap Atrial Fibrillation Group
Number analyzed (Participants) | 0 | 0 | 0

4. Other Pre Specified Outcome: Evaluate the Effect of Cycle Length on Electrogram Duration in Normal Subjects
Description: A change in electrogram duration (in ms) between long and short pacing cycle length.
Time Frame: During ablation procedure
Population: as for baseline characteristics
Arm/Group | Normal Subject Control Group | Atrial Fibrillation Group | AcQMap Atrial Fibrillation Group
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Effect of Pacing Cycle Length on Electrogram Morphology
Description: A change in electrogram morphology from normal to abnormal (defined as ≥3 deflections lasting ≥50ms) between long and short pacing cycle length in regions of low (<0.5mV), intermediate (0.5-lower limit of normal defined from control group) and normal (defined from control group results) voltage amplitude.
Time Frame: During ablation procedure
Reporting Status: Not Posted, anticipated posting 2025-12

6. Secondary Outcome: Effect of Pacing Cycle Length on Conduction Velocity
Description: Difference in single vector conduction velocity at long and short cycle lengths in regions of low, intermediate and normal voltage.
Time Frame: During ablation procedure
Reporting Status: Not Posted, anticipated posting 2025-12

7. Secondary Outcome: To Compare Electroanatomic Voltage Mapping (EAVM) Performed With a Bipolar Contact Force Guided Ablation Catheter to the Abbott HD Grid Using Orthogonal Wave Analysis in Sinus Rhythm.
Description: Difference in voltage amplitude by each method in sinus rhythm.
Time Frame: During ablation procedure
Reporting Status: Not Posted, anticipated posting 2025-12

8. Secondary Outcome: To Evaluate the Distribution of Late Gadolinium Enhancement on Cardiac MRI Relative to Electrogram Amplitude Identified Using the HD Grid
Description: Difference in electrogram voltage amplitude at long and short cycle length in regions with and without late gadolinium enhancement on cardiac MRI.
Time Frame: During ablation procedure
Population: This secondary aim could not be achieved as the cardiac MRI images were too poor to collect measurement values for the pre-specified outcome measure. Therefore, data will never be obtained in the future.
Arm/Group | Normal Subject Control Group | Atrial Fibrillation Group | AcQMap Atrial Fibrillation Group
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: To Evaluate the Distribution of Electrogram Morphologies Relative to Late Gadolinium Enhancement on Cardiac MRI
Description: Difference in proportion of abnormal electrograms >50ms duration and >3 deflections at long and short cycle length in regions with and without late gadolinium enhancement on cardiac MRI.
Time Frame: During ablation procedure
Population: as for outcome 8
Arm/Group | Normal Subject Control Group | Atrial Fibrillation Group | AcQMap Atrial Fibrillation Group
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: To Evaluate the Effect of Cycle Length on Conduction Velocities Relative to Distribution of Late Gadolinium Enhancement on Cardiac MRI
Description: Difference in conduction velocities at long and short cycle length in regions with and without late gadolinium enhancement on cardiac MRI.
Time Frame: During ablation procedure
Population: as for outcome 8
Arm/Group | Normal Subject Control Group | Atrial Fibrillation Group | AcQMap Atrial Fibrillation Group
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Post-procedure assessment on the day of the procedure.
Description: Due to recruitment challenges during the COVID-19 pandemic, we were unable to enroll normal subjects as initially planned.
Arm/Group | Normal Subject Control Group | Atrial Fibrillation Group | AcQMap Atrial Fibrillation Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/18 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/18 | 0/10
Other Adverse Events (participants affected / at risk) | 0/0 | 0/18 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT04229472/Prot_SAP_000.pdf